CLINICAL TRIAL: NCT00993434
Title: The Impact of Educational Materials on Family Behavior
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M-2009-1162
Record Dates: First submitted 2009-10-08; First posted 2009-10-12 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2012-11

CONDITIONS: Overweight; Obesity
Keywords: Child
MeSH Terms: conditions — Overweight; Obesity | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Kid STRIDE Booklet (Active Comparator)
  Interventions: Behavioral: Booklet on nutrition and physical activity.
- Safety Booklet (Placebo Comparator)
  Interventions: Behavioral: Safety Booklet

INTERVENTIONS:
Behavioral: Booklet on nutrition and physical activity. — Parents will be asked to read the booklet and complete a pre- and post-questionnaire.
  Arms: Kid STRIDE Booklet
Behavioral: Safety Booklet — Parents will be asked to read a safety booklet and complete a pre- and post-questionnaire.
  Arms: Safety Booklet

SUMMARY:
The purpose of the research is to learn whether written materials or handouts that are given to parents are helpful in changing knowledge or behavior.

DETAILED DESCRIPTION:
Few written resources for families have been tested in the primary care setting. Kid STRIDE (STRiving to Improve Diet & Exercise) is an educational booklet designed for parents of overweight children. We hypothesize that this booklet will benefit a small percentage of the overweight and obese population of children as a first-tiered approach to treatment of overweight and obese children.

ELIGIBILITY:
Inclusion Criteria:

* Children with a BMI greater than or equal to 85% along with a parent.
* All subjects must speak English.

Exclusion Criteria:

* Genetic conditions associated with overweight.
* Endocrine conditions associated with overweight.
* Chronic steroid therapy.
* Current enrollment in a professional weight management program.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 95 (Actual)
Dates: Start 2009-10; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Assess the effectiveness of written materials on changing knowledge and behavior regarding diet, exercise, and other weight factors. | 3 months

SECONDARY OUTCOMES:
Assess the impact of the intervention on height and weight as reflected in a change in BMI z-score. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Ellen R Wald, MD, Principal Investigator — University of Wisconsin Madison Dept of Pediatrics
Locations (4):
- United States (4):
  - GHC Capitol Pediatric Clinic, Madison, Wisconsin
  - UW Health East Towne Pediatrics, Madison, Wisconsin
  - UW Health West Towne Pediatrics, Madison, Wisconsin
  - UW Health Park Street Pediatrics, Madison, Wisconsin